CLINICAL TRIAL: NCT05016258
Title: Multicenter Observational Study on Performance and Safety Use of "KONTACT MB" Dental Implant in Daily Practice
Brief Title: Performance and Safety Use of the Mono Block Implant "KONTACT MB"
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Biotech Dental (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-A01757-34
Record Dates: First submitted 2021-08-16; First posted 2021-08-23 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-03

CONDITIONS: Dentistry; Dental Implant; Dental Restoration; Implant-supported Fixed Prosthesis
Keywords: Mono Block design; KONTACT MB; Biotech Dental

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- KONTACT MB: Adult patients needed one or multiple implant-supported fixed restoration(s)
  Interventions: Device: KONTACT MB

INTERVENTIONS:
Device: KONTACT MB — Dental implant surgery
  Other Names: Biotech Dental

SUMMARY:
A multicenter prospective observational study aims to illustrate the clinical outcome of dental implants "Kontact MB" and the effects of its Mono Block design on the peri implant bone tissue recession and soft tissue conservation.

All the enrolled patients will be eligible for one or multiple implant-supported fixed restoration(s) according to the routine clinical practice and the manufacturer's instruction for use.

ELIGIBILITY:
Inclusion Criteria:

* Edentulous patient (partially or completely AND formerly, recently or just before implantation) requiring the placement of one (or more) dental implant (s) in maxillary or mandibular
* Age ≥ 18 years
* Good general health (ASA score between [1-2])
* Sufficient bone volume and quality (with or without bone graft) to support the implant
* Given a writing consent for the collection of his medical data as part of the study (delivery of a patient's sheet)

Exclusion Criteria:

* Poor oral hygiene
* Bruxism, parafunctional habits, occlusion disorders and / or temporomandibular joints
* Infections and oral inflammation such as periodontitis, gingivitis
* Patient with metabolic disorders (eg diabetes mellitus) or bone disease that may compromise peri-implant tissue healing
* Heavy smoker (> 10 cigarettes / day)
* Patient with a pathology or immunosuppressive therapy such as chemotherapy, radiotherapy
* Patient on prolonged steroid therapy
* Titanium / titanium alloy allergy
* Alcohol or drug abuse
* Pregnant woman (or likely to be pregnant); or breastfeeding
* Difficulty of medical follow-up patients with geographical, social or psychological constraints
* Persons deprived of liberty or guardianship
* Involuntary / patient refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who is eligible and planned for an implant-supported prosthetic restoration following the instructions for use of the KONTACT MB implant and who meets the inclusion / exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Estimated)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Implant survival rate | up to 36 months
  Number of implants still in function up to 36 months post implantation
Peri implant bone level | up to 36 months
  Bone level evolution compare to the bone level at implantation day
Keratinized tissues level | up to 36 months
  Assessment of keratinized tissues
Gingival index | up to 36 months
  Gingival index assess with Loë and Silness Score
Bleeding index | up to 36 months
  Bleeding index on probing following the Mombelli score

CONTACTS AND LOCATIONS:
Overall Officials: Hadi Antoun, Principal Investigator — Hadi Antoun office
Locations (1):
- Hadi Antoun Office, Paris, France

IPD SHARING:
Plan to Share IPD: No